CLINICAL TRIAL: NCT00140400
Title: Phase I/II Study of a Prime-Boost Schedule of Human GM-CSF Gene Transduced Irradiated Prostate Allogeneic Cancer Vaccine (Allogeneic Prostate GVAX®) in Hormone-Refractory Prostate Cancer
Brief Title: Prime-Boost Dose Scheduling Trial for Human GM-CSF Gene Transduced Irradiated Prostate Allogeneic Cancer Vaccine (Allogeneic Prostate GVAX®) in Patients With Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-9803
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2005-09-01 (Estimated); Status verified 2005-08

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Advanced prostate cancer; Metastatic; Hormone-refractory; GVAX; Vaccine; Allogeneic cells
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Biological: Immunotherapy allogeneic GM-CSF secreting cellular vaccine

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of a prime-boost dose schedule of Human GM-CSF Gene Transduced Irradiated Prostate Allogeneic Cancer Vaccine (Allogeneic Prostate GVAX®) as measured by standard toxicity evaluation, changes in PSA, and tumor responses. Additional objectives are to measure the time to PSA and/or clinical disease progression as well as local and systemic immune responses to the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma prostate cancer
* Prostate cancer deemed to be unresponsive or refractory to hormone therapy
* An ECOG performance status of 0 or 1

Exclusion Criteria:

* Transitional cell, small cell, neuroendocrine, or squamous cell prostate cancer
* Previous chemotherapy, biological or immunotherapy for cancer
* Previous gene therapy for cancer
* Significant cancer related pain

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1999-05; Study Completion 2001-01